CLINICAL TRIAL: NCT05446142
Title: A PHASE 1, RANDOMIZED, OPEN-LABEL STUDY IN HEALTHY PARTICIPANTS TO ESTIMATE THE BIOAVAILABILITY OF TWO NEW ENCORAFENIB FORMULATIONS RELATIVE TO THE CURRENT FORMULATION AND TO EVALUATE THE EFFECT OF A PROTON-PUMP INHIBITOR ON ENCORAFENIB PLASMA PHARMACOKINETICS
Brief Title: A Relative Bioavailability Study Evaluating Two New Encorafenib Formulations
Acronym: ERBA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry); Pierre Fabre Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C4221024
Record Dates: First submitted 2022-07-01; First posted 2022-07-06 (Actual); Results first posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-07

CONDITIONS: Healthy
Keywords: Encorafenib; Rabeprazole; Healthy adult participants
MeSH Terms: interventions — encorafenib; Dosage Forms; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Four Period Treatment Sequence: PPI Effect (Experimental): Participants will receive a single encorafenib dose formulation, a single encorafenib dose of the formulated capsule (CAP), and a single encorafenib dose of the formulation after administration of 20 mg rabeprazole every evening for 5 days.
  Interventions: Drug: Encorafenib capsule formulation (CAP); Drug: Encorafenib first formulation; Drug: Encorafenib second formulation; Drug: Rabeprazole tablet
- Four Period Treatment Sequence: PPI Effect Second Formulation (Experimental): Participants will receive a single encorafenib dose of the second formulation, a single encorafenib dose of the second formulation, a single encorafenib dose of the formulated capsule (CAP), and a single encorafenib dose of the second formulation after administration of 20 mg rabeprazole every evening for 5 days.
  Interventions: Drug: Encorafenib capsule formulation (CAP); Drug: Encorafenib first formulation; Drug: Encorafenib second formulation; Drug: Rabeprazole tablet

INTERVENTIONS:
Drug: Encorafenib capsule formulation (CAP) — A single encorafenib dose of the CAP formulation
Drug: Encorafenib first formulation — first formulation
Drug: Encorafenib second formulation — second formulation
Drug: Rabeprazole tablet — Proton-pump inhibitor

SUMMARY:
Relative bioavailability study to evaluate the pharmacokinetics of two new encorafenib formulations

DETAILED DESCRIPTION:
In order to decrease the size of the current formulated encorafenib capsule and improve the physical stability, 2 new encorafenib tablet formulations have been developed.

This study is intended to select the optimal tablet formulation for commercialization based on the tablet pharmacokinetics.

A preliminary assessment of the effect of a proton-pump inhibitor on the pharmacokinetics of the 2 encorafenib tablet formulations will also be conducted to assist in the formulation selection.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be male or female of non-childbearing potential of 18 years of age or older, inclusive, at the time of signing the informed consent document.
* Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Body Mass Index of 17.5 to 30.5 kg/meters squared; and a body weight >50 kg (110 lb).
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent document and the protocol.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease. Evidence of any active and uncontrolled bacterial or viral infection.
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* History of human immunodeficiency virus infection, hepatitis B, or hepatitis C; positive testing for human immunodeficiency virus, Hepatitis B surface antigen, Hepatitis B core antibody or hepatitis C virus antibody. Hepatitis B vaccination is allowed.
* Positive COVID-19 test at first admission.
* Other medical or psychiatric conditions, laboratory test abnormalities, other conditions or situations related to COVID-19 pandemic or, in the investigator's judgment, make the participant inappropriate for the study.
* Use of prescription or non-prescription medications within 7 days prior to the first dose of encorafenib with the exception of moderate/potent CYP3A inducers which are prohibited within 14 days plus 5 half-lives prior to the first dose.
* History of known sensitivity to rabeprazole, substituted benzimidazoles or to any component of the rabeprazole formulation.
* Previous administration with an investigational product (drug or vaccine) within 30 days.
* Known hypersensitivity to encorafenib or its excipients.
* A positive urine drug or cotinine test.
* Screening supine blood pressure ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest.
* Baseline standard 12 lead electrocardiogram that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results.
* Aspartate transaminase or alanine aminotransferase level ≥ 1.5 × upper limit of normal.
* Total bilirubin level ≥1.5 × upper limit of normal.
* Estimated glomerular filtration rate <60 ml/min/1.73 m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4221024

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 18 participants were enrolled and randomized into 1 of the 6 treatment sequences.
Groups:
- Encorafenib 75 mg eMCC=>75 mg eMCCL=>75 mg CAP=>75 mg eMCC+20 mg Rabeprazole: Period 1: Participants received a single oral dose of encorafenib 75 mg as eMCC under fasted condition, followed by serial PK sampling from Day 1 to Day 3, and a washout of at least 5 days between successive encorafenib dose.
  Period 2: Participants received a single oral dose of encorafenib 75 mg as eMCCL under fasted condition, followed by serial PK sampling from Day 1 to Day 3, and a washout of at least 5 days between successive encorafenib dose.
  Period 3: Participants received a single oral dose of encorafenib 75 mg as CAP under fasted condition, followed by serial PK sampling from Day 1 to Day 3, and a washout of at least 5 days between successive encorafenib dose.
  Period 4: Participants received rabeprazole 20 mg daily from Day -5 to -1, and a single oral dose of encorafenib 75 mg eMCC on Day 1 under fasted condition, followed by serial PK sampling from Day 1 to Day 3.
- Encorafenib 75 mg eMCC=>75 mg CAP=>75 mg eMCCL=>75 mg eMCCL+20 mg Rabeprazole: Period 1: Participants received a single oral dose of encorafenib 75 mg as eMCC under fasted condition, followed by serial PK sampling from Day 1 to Day 3, and a washout of at least 5 days between successive encorafenib dose.
  Period 2: Participants received a single oral dose of encorafenib 75 mg as CAP under fasted condition, followed by serial PK sampling from Day 1 to Day 3, and a washout of at least 5 days between successive encorafenib dose.
  Period 3: Participants received a single oral dose of encorafenib 75 mg as eMCCL under fasted condition, followed by serial PK sampling from Day 1 to Day 3, and a washout of at least 5 days between successive encorafenib dose.
  Period 4: Participants received rabeprazole 20 mg daily from Day -5 to -1, and a single oral dose of encorafenib 75 mg eMCCL on Day 1 under fasted condition, followed by serial PK sampling from Day 1 to Day 3.
- Encorafenib 75 mg eMCCL=>75 mg CAP=>75 mg eMCC=>75 mg eMCC+20 mg Rabeprazole: Period 1: Participants received a single oral dose of encorafenib 75 mg as eMCCL under fasted condition, followed by serial PK sampling from Day 1 to Day 3, and a washout of at least 5 days between successive encorafenib dose.
  Period 2: Participants received a single oral dose of encorafenib 75 mg as CAP under fasted condition, followed by serial PK sampling from Day 1 to Day 3, and a washout of at least 5 days between successive encorafenib dose.
  Period 3: Participants received a single oral dose of encorafenib 75 mg as eMCC under fasted condition, followed by serial PK sampling from Day 1 to Day 3, and a washout of at least 5 days between successive encorafenib dose.
  Period 4: Participants received rabeprazole 20 mg daily from Day -5 to -1, and a single oral dose of encorafenib 75 mg eMCC on Day 1 under fasted condition, followed by serial PK sampling from Day 1 to Day 3.
- Encorafenib 75 mg eMCCL=>75 m eMCC=>75 mg CAP=>75 mg eMCCL+20 mg Rabeprazole: Period 1: Participants received a single oral dose of encorafenib 75 mg as eMCCL under fasted condition, followed by serial PK sampling from Day 1 to Day 3, and a washout of at least 5 days between successive encorafenib dose.
  Period 2: Participants received a single oral dose of encorafenib 75 mg as eMCC under fasted condition, followed by serial PK sampling from Day 1 to Day 3, and a washout of at least 5 days between successive encorafenib dose.
  Period 3: Participants received a single oral dose of encorafenib 75 mg as CAP under fasted condition, followed by serial PK sampling from Day 1 to Day 3, and a washout of at least 5 days between successive encorafenib dose.
  Period 4: Participants received rabeprazole 20 mg daily from Day -5 to -1, and a single oral dose of encorafenib 75 mg eMCCL on Day 1 under fasted condition, followed by serial PK sampling from Day 1 to Day 3.
- Encorafenib 75 mg CAP=>75 mg eMCC=>75 mg eMCCL=>75 mg eMCC+20 mg Rabeprazole: Period 1: Participants received a single oral dose of encorafenib 75 mg as CAP under fasted condition, followed by serial PK sampling from Day 1 to Day 3, and a washout of at least 5 days between successive encorafenib dose.
  Period 2: Participants received a single oral dose of encorafenib 75 mg as eMCC under fasted condition, followed by serial PK sampling from Day 1 to Day 3, and a washout of at least 5 days between successive encorafenib dose.
  Period 3: Participants received a single oral dose of encorafenib 75 mg as eMCCL under fasted condition, followed by serial PK sampling from Day 1 to Day 3, and a washout of at least 5 days between successive encorafenib dose.
  Period 4: Participants received rabeprazole 20 mg daily from Day -5 to -1, and a single oral dose of encorafenib 75 mg eMCC on Day 1 under fasted condition, followed by serial PK sampling from Day 1 to Day 3.
- Encorafenib 75 mg CAP=>75 mg eMCCL=>75 mg eMCC=>75 mg eMCCL+20 mg Rabeprazole: Period 1: Participants received a single oral dose of encorafenib 75 mg as CAP under fasted condition, followed by serial PK sampling from Day 1 to Day 3, and a washout of at least 5 days between successive encorafenib dose.
  Period 2: Participants received a single oral dose of encorafenib 75 mg as eMCCL under fasted condition, followed by serial PK sampling from Day 1 to Day 3, and a washout of at least 5 days between successive encorafenib dose.
  Period 3: Participants received a single oral dose of encorafenib 75 mg as eMCC under fasted condition, followed by serial PK sampling from Day 1 to Day 3, and a washout of at least 5 days between successive encorafenib dose.
  Period 4: Participants received rabeprazole 20 mg daily from Day -5 to -1, and a single oral dose of encorafenib 75 mg eMCCL on Day 1 under fasted condition, followed by serial PK sampling from Day 1 to Day 3.
Period: Period 1
Arm/Group | Encorafenib 75 mg eMCC=>75 mg eMCCL=>75 mg CAP=>75 mg eMCC+20 mg Rabeprazole | Encorafenib 75 mg eMCC=>75 mg CAP=>75 mg eMCCL=>75 mg eMCCL+20 mg Rabeprazole | Encorafenib 75 mg eMCCL=>75 mg CAP=>75 mg eMCC=>75 mg eMCC+20 mg Rabeprazole | Encorafenib 75 mg eMCCL=>75 m eMCC=>75 mg CAP=>75 mg eMCCL+20 mg Rabeprazole | Encorafenib 75 mg CAP=>75 mg eMCC=>75 mg eMCCL=>75 mg eMCC+20 mg Rabeprazole | Encorafenib 75 mg CAP=>75 mg eMCCL=>75 mg eMCC=>75 mg eMCCL+20 mg Rabeprazole
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Encorafenib 75 mg eMCC=>75 mg eMCCL=>75 mg CAP=>75 mg eMCC+20 mg Rabeprazole | Encorafenib 75 mg eMCC=>75 mg CAP=>75 mg eMCCL=>75 mg eMCCL+20 mg Rabeprazole | Encorafenib 75 mg eMCCL=>75 mg CAP=>75 mg eMCC=>75 mg eMCC+20 mg Rabeprazole | Encorafenib 75 mg eMCCL=>75 m eMCC=>75 mg CAP=>75 mg eMCCL+20 mg Rabeprazole | Encorafenib 75 mg CAP=>75 mg eMCC=>75 mg eMCCL=>75 mg eMCC+20 mg Rabeprazole | Encorafenib 75 mg CAP=>75 mg eMCCL=>75 mg eMCC=>75 mg eMCCL+20 mg Rabeprazole
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 2 | 3 | 3 | 3 | 3 | 3
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Encorafenib 75 mg eMCC=>75 mg eMCCL=>75 mg CAP=>75 mg eMCC+20 mg Rabeprazole | Encorafenib 75 mg eMCC=>75 mg CAP=>75 mg eMCCL=>75 mg eMCCL+20 mg Rabeprazole | Encorafenib 75 mg eMCCL=>75 mg CAP=>75 mg eMCC=>75 mg eMCC+20 mg Rabeprazole | Encorafenib 75 mg eMCCL=>75 m eMCC=>75 mg CAP=>75 mg eMCCL+20 mg Rabeprazole | Encorafenib 75 mg CAP=>75 mg eMCC=>75 mg eMCCL=>75 mg eMCC+20 mg Rabeprazole | Encorafenib 75 mg CAP=>75 mg eMCCL=>75 mg eMCC=>75 mg eMCCL+20 mg Rabeprazole
Started | 2 | 3 | 3 | 3 | 3 | 3
Completed | 2 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Encorafenib 75 mg eMCC=>75 mg eMCCL=>75 mg CAP=>75 mg eMCC+20 mg Rabeprazole | Encorafenib 75 mg eMCC=>75 mg CAP=>75 mg eMCCL=>75 mg eMCCL+20 mg Rabeprazole | Encorafenib 75 mg eMCCL=>75 mg CAP=>75 mg eMCC=>75 mg eMCC+20 mg Rabeprazole | Encorafenib 75 mg eMCCL=>75 m eMCC=>75 mg CAP=>75 mg eMCCL+20 mg Rabeprazole | Encorafenib 75 mg CAP=>75 mg eMCC=>75 mg eMCCL=>75 mg eMCC+20 mg Rabeprazole | Encorafenib 75 mg CAP=>75 mg eMCCL=>75 mg eMCC=>75 mg eMCCL+20 mg Rabeprazole
Started | 2 | 3 | 3 | 3 | 3 | 3
Completed | 2 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all enrolled participants.
Groups:
- All Participants: All participants enrolled in this study
Arm/Group | All Participants
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Mean (SD) | 46.5 (15.93)
Age, Customized [Number; unit: Participants]
  18-44 Years | 9
  45-64 Years | 7
  >=65 Years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 13
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 7
  Black or African American | 8
  Asian | 1
  American Indian or Alaska Native | 1
  Black or African American, White | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 13

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to Extrapolated Infinite Time (AUCinf) Following Single Oral Doses of Encorafenib 75 mg Alone and With Rabeprazole
Description: AUCinf for encorafenib eMCC, eMCCL and CAP formulations (75 mg, single dose administration), and for encorafenib eMCC and eMCCL formulations (75 mg, single dose administration) following 5 days of rabeprazole 20 mg daily were calculated by AUClast + (Clast/kel), where AUClast was the area under the plasma concentration-time profile from time zero to last quantifiable concentration, Clast was the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis, and kel was first-order elimination rate constant.
Time Frame: Day 1 predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24, 48 hours postdose
Population: The PK parameter analysis population is defined as all participants randomized and treated who have at least 1 of the encorafenib plasma PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- 75 mg Encorafenib eMCC, Fasted: Participants received a single oral dose of encorafenib 75 mg eMCC under fasted condition.
- 75mg Encorafenib eMCCL, Fasted: Participants received a single oral dose of encorafenib 75 mg eMCCL under fasted condition.
- 75mg Encorafenib CAP, Fasted: Participants received a single oral dose of encorafenib 75 mg CAP under fasted condition.
- 75mg Encorafenib eMCC + 20 mg Rabeprazole, Fasted: Participants received a single oral dose of encorafenib 75 mg eMCC (fasted) following 5 days of rabeprazole 20 mg daily.
- 75mg Encorafenib eMCCL + 20 mg Rabeprazole, Fasted: Participants received a single oral dose of encorafenib 75 mg eMCCL (fasted) following 5 days of rabeprazole 20 mg daily.
Arm/Group | 75 mg Encorafenib eMCC, Fasted | 75mg Encorafenib eMCCL, Fasted | 75mg Encorafenib CAP, Fasted | 75mg Encorafenib eMCC + 20 mg Rabeprazole, Fasted | 75mg Encorafenib eMCCL + 20 mg Rabeprazole, Fasted
Number analyzed (Participants) | 18 | 17 | 17 | 7 | 9
ng*hr/mL | 2895 (44) | 2909 (49) | 2957 (41) | 2825 (35) | 2556 (63)
Statistical Analysis 1: Comparison: 75 mg Encorafenib eMCC, Fasted vs 75mg Encorafenib CAP, Fasted; Natural log transformed encorafenib AUCinf was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences (eMCC relative to CAP) and corresponding 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (eMCC relative to CAP) and 90% CIs for the ratios. The geometric mean ratios are presented as percentages; Test type: Other; Reference/Test Ratio = 95.25, 90% CI 2-sided [90.82 to 99.90]
Statistical Analysis 2: Comparison: 75mg Encorafenib eMCCL, Fasted vs 75mg Encorafenib CAP, Fasted; Natural log transformed encorafenib AUCinf was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences (eMCCL relative to CAP) and corresponding 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (eMCCL relative to CAP) and 90% CIs for the ratios. The geometric mean ratios are presented as percentages; Test type: Other; Reference/Test Ratio = 96.30, 90% CI 2-sided [91.71 to 101.12]
Statistical Analysis 3: Comparison: 75 mg Encorafenib eMCC, Fasted vs 75mg Encorafenib eMCC + 20 mg Rabeprazole, Fasted; Natural log transformed encorafenib AUCinf was analyzed using ANOVA with treatment and sequence as a fixed effect and participant within sequence as a random effect. The adjusted mean differences (eMCC relative to eMCC with rabeprazole) and corresponding 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (eMCC relative to eMCC with rabeprazole) and 90% CIs for the ratios. The geometric mean ratios are presented as percentages; Test type: Other; Reference/Test Ratio = 96.57, 90% CI 2-sided [82.91 to 112.47]
Statistical Analysis 4: Comparison: 75mg Encorafenib eMCCL, Fasted vs 75mg Encorafenib eMCCL + 20 mg Rabeprazole, Fasted; Natural log transformed encorafenib AUCinf was analyzed using ANOVA with treatment and sequence as a fixed effect and participant within sequence as a random effect. The adjusted mean differences (eMCCL relative to eMCCL with rabeprazole) and corresponding 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (eMCCL relative to eMCCL with rabeprazole) and 90% CIs for the ratios. The geometric mean ratios are presented as percentages; Test type: Other; Reference/Test Ratio = 88.56, 90% CI 2-sided [82.59 to 94.95]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) Following Single Oral Doses of Encorafenib 75 mg Alone and With Rabeprazole
Description: Cmax for encorafenib eMCC, eMCCL and CAP formulations (75 mg, single dose administration), and for encorafenib eMCC and eMCCL formulations (75 mg, single dose administration) following 5 days of rabeprazole 20 mg daily were observed directly from data.
Time Frame: Day 1 predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24, 48 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 75 mg Encorafenib eMCC, Fasted | 75mg Encorafenib eMCCL, Fasted | 75mg Encorafenib CAP, Fasted | 75mg Encorafenib eMCC + 20 mg Rabeprazole, Fasted | 75mg Encorafenib eMCCL + 20 mg Rabeprazole, Fasted
Number analyzed (Participants) | 18 | 18 | 17 | 8 | 9
ng/mL | 898.4 (46) | 778.2 (45) | 845.8 (36) | 686.0 (43) | 631.7 (70)
Statistical Analysis 1: Comparison: 75 mg Encorafenib eMCC, Fasted vs 75mg Encorafenib CAP, Fasted; Natural log transformed encorafenib Cmax was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences (eMCC relative to CAP) and corresponding 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (eMCC relative to CAP) and 90% CIs for the ratios. The geometric mean ratios are presented as percentages; Test type: Other; Reference/Test Ratio = 104.31, 90% CI 2-sided [91.40 to 119.04]
Statistical Analysis 2: Comparison: 75mg Encorafenib eMCCL, Fasted vs 75mg Encorafenib CAP, Fasted; Natural log transformed encorafenib Cmax was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences (eMCCL relative to CAP) and corresponding 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (eMCCL relative to CAP) and 90% CIs for the ratios. The geometric mean ratios are presented as percentages; Test type: Other; Reference/Test Ratio = 90.35, 90% CI 2-sided [79.17 to 103.12]
Statistical Analysis 3: Comparison: 75 mg Encorafenib eMCC, Fasted vs 75mg Encorafenib eMCC + 20 mg Rabeprazole, Fasted; Natural log transformed encorafenib Cmax was analyzed using ANOVA with treatment and sequence as a fixed effect and participant within sequence as a random effect. The adjusted mean differences (eMCC relative to eMCC with rabeprazole) and corresponding 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (eMCC relative to eMCC with rabeprazole) and 90% CIs for the ratios. The geometric mean ratios are presented as percentages; Test type: Other; Reference/Test Ratio = 79.66, 90% CI 2-sided [58.70 to 108.08]
Statistical Analysis 4: Comparison: 75mg Encorafenib eMCCL, Fasted vs 75mg Encorafenib eMCCL + 20 mg Rabeprazole, Fasted; Natural log transformed encorafenib Cmax was analyzed using ANOVA with treatment and sequence as a fixed effect and participant within sequence as a random effect. The adjusted mean differences (eMCCL relative to eMCCL with rabeprazole) and corresponding 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (eMCCL relative to eMCCL with rabeprazole) and 90% CIs for the ratios. The geometric mean ratios are presented as percentages; Test type: Other; Reference/Test Ratio = 80.78, 90% CI 2-sided [64.82 to 100.68]

3. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to Last Quantifiable Concentration (AUClast) Following Single Oral Doses of Encorafenib 75 mg Alone and With Rabeprazole
Description: AUClast for encorafenib eMCC, eMCCL and CAP formulations (75 mg, single dose administration), and for encorafenib eMCC and eMCCL formulations (75 mg, single dose administration) following 5 days of rabeprazole 20 mg daily were calculated using Linear/Log trapezoidal method.
Time Frame: Day 1 predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24, 48 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | 75 mg Encorafenib eMCC, Fasted | 75mg Encorafenib eMCCL, Fasted | 75mg Encorafenib CAP, Fasted | 75mg Encorafenib eMCC + 20 mg Rabeprazole, Fasted | 75mg Encorafenib eMCCL + 20 mg Rabeprazole, Fasted
Number analyzed (Participants) | 18 | 18 | 17 | 8 | 9
ng*hr/mL | 2879 (44) | 2858 (48) | 2934 (41) | 2635 (37) | 2529 (65)
Statistical Analysis 1: Comparison: 75 mg Encorafenib eMCC, Fasted vs 75mg Encorafenib CAP, Fasted; Natural log transformed encorafenib AUClast was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences (eMCC relative to CAP) and corresponding 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (eMCC relative to CAP) and 90% CIs for the ratios. The geometric mean ratios are presented as percentages; Test type: Other; Reference/Test Ratio = 95.34, 90% CI 2-sided [90.37 to 100.59]
Statistical Analysis 2: Comparison: 75mg Encorafenib eMCCL, Fasted vs 75mg Encorafenib CAP, Fasted; Natural log transformed encorafenib AUClast was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences (eMCCL relative to CAP) and corresponding 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (eMCCL relative to CAP) and 90% CIs for the ratios. The geometric mean ratios are presented as percentages; Test type: Other; Reference/Test Ratio = 94.67, 90% CI 2-sided [89.73 to 99.88]
Statistical Analysis 3: Comparison: 75 mg Encorafenib eMCC, Fasted vs 75mg Encorafenib eMCC + 20 mg Rabeprazole, Fasted; Natural log transformed encorafenib AUClast was analyzed using ANOVA with treatment and sequence as a fixed effect and participant within sequence as a random effect. The adjusted mean differences (eMCC relative to eMCC with rabeprazole) and corresponding 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (eMCC relative to eMCC with rabeprazole) and 90% CIs for the ratios. The geometric mean ratios are presented as percentages; Test type: Other; Reference/Test Ratio = 95.76, 90% CI 2-sided [84.10 to 109.04]
Statistical Analysis 4: Comparison: 75mg Encorafenib eMCCL, Fasted vs 75mg Encorafenib eMCCL + 20 mg Rabeprazole, Fasted; Natural log transformed encorafenib AUClast was analyzed using ANOVA with treatment and sequence as a fixed effect and participant within sequence as a random effect. The adjusted mean differences (eMCCL relative to eMCCL with rabeprazole) and corresponding 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (eMCCL relative to eMCCL with rabeprazole) and 90% CIs for the ratios. The geometric mean ratios are presented as percentages; Test type: Other; Reference/Test Ratio = 88.31, 90% CI 2-sided [82.36 to 94.70]

4. Secondary Outcome: Time for Cmax (Tmax) Following Single Oral Doses of Encorafenib 75 mg Alone and With Rabeprazole
Description: Tmax for encorafenib eMCC, eMCCL and CAP formulations (75 mg, single dose administration), and for encorafenib eMCC and eMCCL formulations (75 mg, single dose administration) following 5 days of rabeprazole 20 mg daily were observed directly from data as time of first occurrence.
Time Frame: Day 1 predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24, 48 hours postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | 75 mg Encorafenib eMCC, Fasted | 75mg Encorafenib eMCCL, Fasted | 75mg Encorafenib CAP, Fasted | 75mg Encorafenib eMCC + 20 mg Rabeprazole, Fasted | 75mg Encorafenib eMCCL + 20 mg Rabeprazole, Fasted
Number analyzed (Participants) | 18 | 18 | 17 | 8 | 9
hr | 1.00 [0.500 to 3.00] | 1.00 [1.00 to 1.50] | 1.5 [1.00 to 3.00] | 1.25 [1.00 to 2.52] | 1.00 [0.500 to 3.00]

5. Secondary Outcome: Terminal Half-Life (t½) Following Single Oral Doses of Encorafenib 75 mg Alone and With Rabeprazole
Description: t½ for encorafenib eMCC, eMCCL and CAP formulations (75 mg, single dose administration), and for encorafenib eMCC and eMCCL formulations (75 mg, single dose administration) following 5 days of rabeprazole 20 mg daily were calculated by Loge(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration time curve.
Time Frame: Day 1 predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24, 48 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | 75 mg Encorafenib eMCC, Fasted | 75mg Encorafenib eMCCL, Fasted | 75mg Encorafenib CAP, Fasted | 75mg Encorafenib eMCC + 20 mg Rabeprazole, Fasted | 75mg Encorafenib eMCCL + 20 mg Rabeprazole, Fasted
Number analyzed (Participants) | 18 | 17 | 17 | 7 | 9
hour | 4.691 (1.5680) | 4.850 (2.0588) | 4.730 (1.7416) | 4.710 (2.3714) | 5.350 (2.0893)

6. Secondary Outcome: Apparent Clearance (CL/F) Following Single Oral Doses of Encorafenib 75 mg Alone and With Rabeprazole
Description: CL/F for encorafenib eMCC, eMCCL and CAP formulations (75 mg, single dose administration), and for encorafenib eMCC and eMCCL formulations (75 mg, single dose administration) following 5 days of rabeprazole 20 mg daily were calculated by Dose/AUCinf after oral dose.
Time Frame: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24, 48 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | 75 mg Encorafenib eMCC, Fasted | 75mg Encorafenib eMCCL, Fasted | 75mg Encorafenib CAP, Fasted | 75mg Encorafenib eMCC + 20 mg Rabeprazole, Fasted | 75mg Encorafenib eMCCL + 20 mg Rabeprazole, Fasted
Number analyzed (Participants) | 18 | 17 | 17 | 7 | 9
L/hr | 25.91 (44) | 25.81 (49) | 25.38 (41) | 26.53 (34) | 29.34 (64)

7. Secondary Outcome: Apparent Volume of Distribution (Vz/F) Following Single Oral Doses of Encorafenib 75 mg Alone and With Rabeprazole
Description: Vz/F for encorafenib eMCC, eMCCL and CAP formulations (75 mg, single dose administration), and for encorafenib eMCC and eMCCL formulations (75 mg, single dose administration) following 5 days of rabeprazole 20 mg daily were calculated by Dose/(AUCinf * kel) after oral dose.
Time Frame: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24, 48 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | 75 mg Encorafenib eMCC, Fasted | 75mg Encorafenib eMCCL, Fasted | 75mg Encorafenib CAP, Fasted | 75mg Encorafenib eMCC + 20 mg Rabeprazole, Fasted | 75mg Encorafenib eMCCL + 20 mg Rabeprazole, Fasted
Number analyzed (Participants) | 18 | 17 | 17 | 7 | 9
Liters | 166.1 (46) | 165.1 (49) | 161.7 (46) | 159.3 (29) | 209 (56)

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An serious adverse event (SAE) was defined as an AE: 1. resulting in death, 2. was life-threatening, 3. required inpatient hospitalization or prolongation of existing hospitalization, 4. resulted in persistent disability, 5. was a congenital anomaly/birth defect, or considered to be an important medical event. Any AEs occurring following start of treatment were considered as treatment emergent adverse event (TEAE). Events that occurred during follow-up within the lag time of up to 28 days after the last encorafenib dose were counted as treatment emergent and attributed to the last treatment taken. Events that occurred during the washout period (up to 28 days from the last treatment) between study periods were counted as treatment emergent and attributed to the previous treatment taken.
Time Frame: Baseline up to Day 28 after the last encorafenib dose (the total duration of the study was approximately 60 days from baseline)
Population: All participants randomly assigned to a treatment sequence and who took at least 1 dose of encorafenib. Participants were analyzed according to the formulation they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | 75 mg Encorafenib eMCC, Fasted | 75mg Encorafenib eMCCL, Fasted | 75mg Encorafenib CAP, Fasted | 75mg Encorafenib eMCC + 20 mg Rabeprazole, Fasted | 75mg Encorafenib eMCCL + 20 mg Rabeprazole, Fasted
Number analyzed (Participants) | 18 | 18 | 17 | 8 | 9
Participants
  Participants with AEs (All Causalities) | 11 | 11 | 8 | 1 | 5
  Participants with AEs (Treatment related) | 11 | 9 | 8 | 1 | 5
  Participants with SAEs (All Causalities) | 0 | 0 | 0 | 0 | 0
  Participants with severe (including fatal) adverse events (All Causalities) | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities Without Regard to Baseline Abnormality
Description: Haematological, clinical chemistry (serum) and urinalysis safety tests were assessed against the criteria specified in the sponsor reporting standards. The assessment did not take into account whether each participants's baseline test result was within or outside the laboratory reference range for the particular laboratory parameter. The baseline measurement for safety laboratory tests for all periods was the predose measurement on Day -1 of Period 1. Only those categories in which at least 1 participant had data were reported.
Time Frame: Baseline, and at early discontinuation or at the discretion of the investigator (the total duration of the study was approximately 60 days from baseline)
Population: All participants randomly assigned to a treatment sequence and who took at least 1 dose of encorafenib. Participants were analyzed according to the formulation they actually received. Specifically, number of participants analyzed in the table is the total number of participants with at least one observation of the given laboratory test while on study treatment or during lag time.
Measure: Count of Participants; unit: Participants
Arm/Group | 75 mg Encorafenib eMCC, Fasted | 75mg Encorafenib eMCCL, Fasted | 75mg Encorafenib CAP, Fasted | 75mg Encorafenib eMCC + 20 mg Rabeprazole, Fasted | 75mg Encorafenib eMCCL + 20 mg Rabeprazole, Fasted
Number analyzed (Participants) | 0 | 1 | 0 | 8 | 9
Participants
  HEMATOLOGY - Monocytes/Leukocytes (%) > 1.2 x Upper Limit of Normal (ULN) | 0 | 0 | 0 | 3 | 0
  CLINICAL CHEMISTRY - Urate (mg/dL) > 1.2x ULN | 0 | 0 | 0 | 1 | 0
  URINALYSIS - Urobilinogen (EU) >= 1 | 0 | 0 | 0 | 0 | 1

10. Secondary Outcome: Number of Participants Meeting Vital Signs Categorical Criteria
Description: Supine blood pressure (BP) and pulse rate (PR) were measured at times specified. For Periods 1 to 3, the baseline measurement was the predose measurement on Day -1 of each period. For Period 4, the baseline measurement was the predose measurement on Day -1 of Period 3. The reported categories included: systolic blood pressure (SBP)>=90mmHg; change from baseline (CFB) in SBP>=30mmHg; diastolic blood pressure (DBP)<50mmHg; CFB in DBP>=20mmHg; PR<40 beats per minute (bpm) or PR>120bpm. Only those categories in which at least 1 participant had data were provided.
Time Frame: Baseline, 0 and 2 hours postdose in each period, and at early discontinuation (the total duration of the study was approximately 60 days from baseline)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | 75 mg Encorafenib eMCC, Fasted | 75mg Encorafenib eMCCL, Fasted | 75mg Encorafenib CAP, Fasted | 75mg Encorafenib eMCC + 20 mg Rabeprazole, Fasted | 75mg Encorafenib eMCCL + 20 mg Rabeprazole, Fasted
Number analyzed (Participants) | 18 | 18 | 17 | 8 | 9
Participants | 1 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participnts With Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Absolute values and changes from baseline in PR, QT, QRS, heart rate and QTcF were summarized by protocol pre-defined categorization criterion. QTcF were derived using Fridericia's heart rate correction formula. For each period, triplicate ECGs were conducted predose on Day 1; all other ECG measurements were single ECGs. The baseline ECG value was the average of the triplicate ECG measurements collected before dose administration on Day 1. Changes from baseline were defined as the change between the postdose ECG measurement and the derived baseline ECG.
Time Frame: as for outcome 10
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | 75 mg Encorafenib eMCC, Fasted | 75mg Encorafenib eMCCL, Fasted | 75mg Encorafenib CAP, Fasted | 75mg Encorafenib eMCC + 20 mg Rabeprazole, Fasted | 75mg Encorafenib eMCCL + 20 mg Rabeprazole, Fasted
Number analyzed (Participants) | 18 | 18 | 17 | 8 | 9
Participants
  PR INTERVAL (MSEC) value >= 300 msec or %Chg>=25/50% | 0 | 0 | 0 | 0 | 0
  QRS COMPLEX (MSEC) Value >=140 msec or %Chg>=50% | 0 | 0 | 0 | 0 | 0
  QT INTERVAL (MSEC) Value >=500 msec | 0 | 0 | 0 | 0 | 0
  QTCF (MSEC) 450 msec <= Value < 480 msec or 480 msec <= Value < 500 msec or Value > 500 msec | 0 | 0 | 0 | 0 | 0
  QTCF (MSEC) 30 msec <= Chg < 60 msec or Chg > 60 msec | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Day 28 after the last encorafenib dose. The total duration of the study was approximately 60 days from baseline.
Groups:
- 75 mg Encorafenib eMCC, Fasted: Participants received a single ora l dose of encorafenib 75 mg eMCC under fasted condition.
- 75 mg Encorafenib eMCCL, Fasted: Participants received a single oral dose of encorafenib 75 mg eMCCL under fasted condition.
- 75 mg Encorafenib CAP, Fasted: Participants received a single oral dose of encorafenib 75 mg CAP under fasted condition.
Arm/Group | 75 mg Encorafenib eMCC, Fasted | 75 mg Encorafenib eMCCL, Fasted | 75 mg Encorafenib CAP, Fasted | 75mg Encorafenib eMCC + 20 mg Rabeprazole, Fasted | 75mg Encorafenib eMCCL + 20 mg Rabeprazole, Fasted
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/17 | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/17 | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 11/18 | 11/18 | 8/17 | 1/8 | 5/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 75 mg Encorafenib eMCC, Fasted (N=18) | 75 mg Encorafenib eMCCL, Fasted (N=18) | 75 mg Encorafenib CAP, Fasted (N=17) | 75mg Encorafenib eMCC + 20 mg Rabeprazole, Fasted (N=8) | 75mg Encorafenib eMCCL + 20 mg Rabeprazole, Fasted (N=9)
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Change of bowel habit (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 1
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 2 | 0 | 0 | 0
Feeling hot (General disorders) | 4 | 4 | 1 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 2 | 1 | 0 | 1
Headache (Nervous system disorders) | 4 | 2 | 5 | 1 | 2
Paraesthesia (Nervous system disorders) | 0 | 2 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pseudofolliculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 2 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT05446142/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-04): https://cdn.clinicaltrials.gov/large-docs/42/NCT05446142/SAP_001.pdf